CLINICAL TRIAL: NCT04512872
Title: A Pilot Phase 1, Double-Blind, Randomized, Two-arm, Parallel Group, Single-dose Study to Evaluate the Safety and Pharmacokinetics of CT-P41 and EU-approved Prolia in Healthy Male Subjects
Brief Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of CT-P41 and EU-approved Prolia in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P41 1.1
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P41 (Experimental): 60 mg/mL single dose administration, Solution for injection in PFS
  Interventions: Biological: CT-P41
- EU-approved Prolia (Active Comparator): 60 mg/mL single dose administration, Solution for injection in PFS
  Interventions: Biological: EU-approved Prolia

INTERVENTIONS:
Biological: CT-P41 — 60 mg/mL single dose, Solution for injection in PFS
  Arms: CT-P41
Biological: EU-approved Prolia — 60 mg/mL single dose, Solution for injection in PFS
  Arms: EU-approved Prolia

SUMMARY:
This study is a Pilot Phase 1, Double-Blind, Randomized, Two-arm, Parallel group, Single-dose Study to Evaluate the Safety and Pharmacokinetics of CT-P41 and EU-approved Prolia in Healthy Male Subjects

DETAILED DESCRIPTION:
This study is a pilot phase 1, randomized, double-blind, two-arm, parallel group, single-dose study, which is designed to evaluate the safety, immunogenicity, PK and PD of CT-P41 and EU-approved Prolia in healthy male subjects. Approximately 30 male subjects will be enrolled and randomly assigned to one of the two treatment arms in a 1:1 ratio. In each treatment group, all subjects will receive a single 60 mg dose of either CT P41 or EU-approved Prolia by subcutaneous injection via a PFS on Day 1, followed by 134 days of safety, immunogenicity, PK, and PD measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, between the ages of 28 and 55 years.
* Subject with a BMI between 18.5 and 29.9 kg/m2.
* Subject with albumin-adjusted total serum calcium ≥8.5 mg/dL (≥2.125 mol/L) and serum 25-OH vitamin D ≥20 ng/ml.
* Male subject and their female partner of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 5 months after the study drug administration.

Exclusion Criteria:

* Subject with a hypersensitivity to any component of denosumab.
* Subject has a history of and/or current known risk factors for hypocalcemia and osteonecrosis of jaw, and any clinically significant illness at investigator's discretion.
* Subject has a history of and/or concurrent use of medications such as an investigational drug, monoclonal antibody, fusion protein, and biologics.
* Subject has a history of and/or concurrent use of any therapy that might significantly affect bone metabolism.
* Subject is vulnerable.
* Subject is not likely to complete the study for whatever reason in the opinion of the Investigator.

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Evaluate safety | through study completion, up to day 134
  safety in terms of treatment-emergent adverse events (TEAEs) of CT-P41 compared to that of EU-approved Prolia

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Ltd, Herston, Queensland, Australia